CLINICAL TRIAL: NCT06176950
Title: History of Neonatology
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Johanna Schoen, PhD, Professor of History, Rutgers, The State University of New Jersey
Other Study IDs: Pro2021000877
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Oral History
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Oral History Interviews — I will ask interview subjects about their educational and career path, their research interests and clinical work in the field of neonatology. I will also ask them about their personal and professional motivations and thoughts about their work. And we will discuss how their interactions with colleagues and patients/caregivers shaped their work experience and decision making.

SUMMARY:
This study traces the history of neonatology in the United States from the 1960s to the present with particular attention to the ways in which neonatologists developed criteria to make treatment decisions. I will be using oral history interviews as one source for a book that will document developments in the history of neonatology. I will identify potential research subjects through their publications in the field of neonatology and through word of mouth. I will locate them via the contact information provided in their publications or through an internet search.

DETAILED DESCRIPTION:
I will interview individuals who have worked in NICUs [neonatologists, nurses, social workers] to understand how technological changes and changing scientific understanding influenced decision making pertaining to the treatment of infants. The interviews will supplement my extensive research of the medical literature and other pertinent publications.

Between the 1960s and the present, we have seen the emergence of medical therapies and technologies developed to treat neonates. Over this time period, there has also been a changing and growing understanding of the long-term impact that medical interventions have on the infants treated as well as on their families. Finally, the demographic characteristics of neonates have also changed as public health crises as well as the development of modern reproductive technologies led to new patient populations and new expectations of what NICUs should or should not achieve. I am interested in the ways in which these changes have led to evolving treatment criteria for neonates and ways in which neonatologists decided when to treat and when treatment was considered futile. I will interview medical professionals who are working or have worked at NICUs about the changes they experienced in their place of work over the course of their careers, the impact that medical technologies and changing patient populations had on considerations about treatment options, and the discussions they had with colleagues and the parents of patients.

There is to date no sustained historical analysis of neonatology. There are anthropological studies of the development of fetal surgery [Casper 1998] as well as Assisted Reproductive Technologies [Spar, 2006; Thompson, 2005]. There are analyses of the social history of particular medical interventions [abortion, birth control, etc.] [Schoen, 1995; Schoen 2005] and the treatment of the fetus [Withycombe, 2019]. And scholars have discussed the value of reproduction and the fetus as it pertains to emerging technologies of genetic testing and the history of disability [Davis, 2019; Herzog, 2018; Lowy, 2018; Maienschein, 2003; Maienschein, 2014; Rapp, 2000; Reagan, 2010.] This study will contribute to our understanding of the ways in which medical professionals have made decisions about life, death, and the quality of life of those being treated.

ELIGIBILITY:
Inclusion Criteria: I will interview individuals who worked or are working in Neonatal Intensive Care Units as neonatologists, pediatricians, nurses, social workers or other pertinent professionals in the medical or counseling field.

Exclusion Criteria: N/A

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: individuals who have worked in NICUs [neonatologists, nurses, social workers] in the 20th and/or early 21st century
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Information about the history of neonatology | 2 hours
  Interviews will be transcribed and indexed by key words pertaining to the history of NICUs

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Schoen, PhD, Principal Investigator — Johanna Schoen
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
If interview subjects agree, I will donate the interviews to the American Academia of Pediatrics which has an archive of oral histories with pediatricians and neonatologists.
Supporting Information: Study Protocol, ICF
Time Frame: December 2028 anticipated
Access Criteria: anyone who wishes to access the data